CLINICAL TRIAL: NCT06092762
Title: a Multicenter, Randomized, Open Label Phase II Clinical Study to Evaluate the Safety and Efficacy of AK120 in the Treatment of Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety and Efficacy of AK120 in Subjects With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK120-206
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK120 300mg (Experimental): AK120 loading dose 600mg, then 300mg subcutaneous injection every 2 weeks thereafter until week 14.
  Interventions: Drug: AK120
- AK120 450mg (Experimental): AK120 loading dose 600mg, then 450mg subcutaneous injection every 2 weeks thereafter until week 14.
  Interventions: Drug: AK120

INTERVENTIONS:
Drug: AK120 — subcutaneous injection every 2 weeks

SUMMARY:
This is a multicenter, randomized, open label phase II clinical study to evaluate the safety and efficacy of AK120 in the treatment of subjects with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open label phase II clinical study to evaluate the safety and efficacy of AK120 in the treatment of subjects with moderate to severe atopic dermatitis. The total duration of the study (including screening period) planned for each subject is approximately 29 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18≤75 years old.
2. Atopic dermatitis (AD) diagnosed at least half a year before screening.
3. Subject with EASI score ≥16, IGA ≥ 3, BSA ≥ 10% at screening and baseline.
4. Subjects with a history of an inadequate response or medically inappropriate use of topical drug treatment within 6 months

Exclusion Criteria:

1. Received systemic corticosteroids, immunosuppressive/immunomodulatory drugs, phototherapy within the 4 weeks before randomization.
2. Received systemic traditional Chinese medicine treatment within the 4 weeks before randomization or topical traditional Chinese medicine treatment within 1 week before randomization
3. Received treatment with other clinical study drugs within 1 month or 5 half-lives before randomization (whichever is longer)
4. Received or planned to receive live vaccine treatment within the 3 months before randomization or during the study period.
5. Received allergen specific immunotherapy within the 3 months before randomization.
6. Have a history of allergies to any component of AK120 and/or severe allergic reactions to monoclonal antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) | week 0 to week 24
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment

SECONDARY OUTCOMES:
Percentage of subjects who achieved (Eczema Area and Severity Index) EASI-75 | at week 2/4/8/12/16 /20 and 24
Percentage of subjects who achieved (Eczema Area and Severity Index) EASI-50 | at week 2/4/8/12/16 /20 and 24
Percentage change in (Eczema Area and Severity Index) EASI scores from baseline | at week 2/4/8/12/16 /20 and 24
Percentage of subjects who achieved 0/1 in the (Investigator's Global Assessment) IGA | at week 2/4/8/12/16 /20 and 24
Percentage of subjects with a (Investigator's Global Assessment) IGA score decrease of ≥ 2 points from baseline | at week 2/4/8/12/16 /20 and 24
Percentage change in (affected body surface area) BSA score from baseline | at week 2/4/8/12/16 /20 and 24

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Air Force Medical Center, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Xiamen Medical College, Xiamen, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - People Hospital of Xingtai, Xingtai, Hebei
  - Renmin Hospital of Wuhan University Hubei General Hospital, Wuhan, Hubei
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Yancheng No.1 People's Hospital, Yancheng, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Baoji Central Hospital, Baoji, Shanxi
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Taiyuan Central Hospital, Taiyuan, Shanxi
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital，Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang
  - The first affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang

IPD SHARING:
Plan to Share IPD: No